CLINICAL TRIAL: NCT06788379
Title: CENP-V As a Potential Diagnostic Marker of Damage in Human Oocytes
Acronym: CENP-PILOT
Status: Recruiting | Type: Observational
Sponsor: Vida Recoletas Sevilla (Other)
Collaborators: University of Seville, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-SEV-102-MF
Record Dates: First submitted 2024-10-04; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Establish the Amount of CENPV Protein in Human Oocytes As a Diagnostic Tool Against Damage Caused by Ageing or by the Procedure of Vitrification of Oocytes; Advance Maternal Age; Vitrification and Thawing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Patients with advanced maternal age (AMA): Patients aged 36-45 years with AMA etiology as the main factor of infertility undergoing controlled ovarian stimulation
- Control patients: Patients and donors with normal etiology, aged 18-35 years, undergoing controlled ovarian stimulation and collection procedures.

SUMMARY:
Proper chromosome segregation is essential to avoid aneuploidy, yet in mammalian oocytes it progressively fails in an age-dependent manner. The ageing population and the increasing age of parenthood are leading to a declined fertility. Proteins contributing to correct chromosome segregation and oocyte ageing are therefore of central interest. Mouse oocytes deficient in CENP-V are strongly impaired in meiosis I. The spindle assembly checkpoint (SAC)-dependent arrest of about half of the Cenp-V -/- oocytes at metaphase I is only found in oocytes from young adults, not in oocytes >12 months. This suggests SAC weakening in ageing oocytes allowing them to proceed despite continuous presence of mis-aligned chromosomes and present CENP-V depleted oocytes as a model for age dependent weakening of the SAC. Sporadic cases of very-low oocyte survival rate have been observed after vitrification and thawing protocols in the clinical practice. However, no diagnostic tools are currently available to detect these cases. The relevance of this problem has led to a demand on the scientific community to obtain specific and early biomarkers to predict decreased oocyte survival rates after thawing. The main goal of this project is to establish the expression levels of the CENP-V protein in human oocytes as a diagnostic tool for the aging of a cohort of oocytes. With this purpose, the immature oocytes from the oocytes cohort recovered from women with advanced maternal age (AMA) and control, will be matured in vitro in order to compare the CENP-V expression levels between both populations. In addition, in patients with AMA, these expression levels will be correlated with the aneuploidy rate from the blastocyst of the same oocyte cohort. CENP-V-deleted mouse oocytes show higher rate of aneuploidy and spindle aberrations after cold treatment compared to control oocytes. We hypothesize that alterations in the expression level of CENP-V could be responsible of the decrease in oocyte survival rate after thawing. The main objective of this project is to establish the expression levels of the CENP-V protein in human oocytes as a diagnostic tool to assess the damage of a cohort of oocytes. For this purpose, oocytes retrieved from advanced maternal age (AMA) and control patients, as well as oocytes undergoing vitrification / thawing procedures and controls oocytes, will be analyzed. In this study, only the immature oocytes of the patients, which are destined to be discarded and not used in their treatment, will be analyzed.

DETAILED DESCRIPTION:
This is a prospective, unicentric, descriptive and transversal study. The main objective of this project is to establish the expression levels of the CENP-V protein in human oocytes as a diagnostic tool of damage in a cohort of human oocytes. With this purpose, CENP-V levels of discarded oocytes retrieved from Advanced Maternal Age (AMA) and control patients will be analyzed in fresh state and after vitrification-thawing procedures. As mature oocytes will be used for the patient's treatment, only immature oocytes, that would otherwise have been discarded, or mature oocyte donated to research, will be used in this project.

ELIGIBILITY:
Inclusion Criteria:

* Group of patients with advanced maternal age (AMA): patients aged 36-45 years with AMA etiology as the main factor of infertility undergoing controlled ovarian stimulation.
* Group of patients with vitrification / thawing of their oocytes: patients between 18-45 years of age who underwent oocyte vitrification to later, in the study cycle, thaw their oocytes. In this group we contemplate two subgroups:

  * Patients with vitrified / thawed oocytes and AMA: between 36-45 years at the moment of oocytes vitrification.
  * Patients with vitrified / thawed oocytes and non-AMA: between 18-35 years at the moment of oocytes vitrification.
* Group of control patients: patients and donors with normal etiology, aged 18-35 years, undergoing controlled ovarian stimulation and collection procedures.

Exclusion Criteria:

* Patients with pathologies affecting the oocyte quality (PCO, POI, endometriosis, oncology patients, etc.).
* Patients/donors with oocyte cryopreserved by slow freezing technique.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The reference population will be constituted of patients and donors with immature oocytes(GV, MI), obtained after oocyte collection, and mature oocytes (MII) vitrified from patients who decide not to use them and are willing to donate them to research projects. Women willing to participate in this study will be previously informed and will have to sign the informed consent form of the study. The recruitment of patients will be performed in IVI RMA Seville clinic.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CENP-V levels y distribution in oocyte | From enrollment to oocyte retrieval, two days

SECONDARY OUTCOMES:
Survival rate of the oocyte cohort | From enrollment to oocyte retrieval, two days

CONTACTS AND LOCATIONS:
Locations (1):
- Vida Recoletas Sevilla S.L., Seville, SEVILLA, Spain